CLINICAL TRIAL: NCT01283867
Title: An Open-label, Balanced, Randomized, Two-treatment, Two-period, Two Sequence, Single Dose, Crossover, Bioequivalence Study of Mycophenolate Mofetil 500 mg Tablet of Dr. Reddy's Laboratories Limited Comparing With That of Cellcept 500 mg Tablet of Roche Laboratories in Healthy, Adult,Human, Male Subjects Under Non-fasting Conditions.
Brief Title: Bioequivalence Study of Mycophenolate Mofetil 500 mg Tablets of Dr.Reddy's Laboratories Limited Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Director-Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 295-07
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: FED
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mycophenolate Mofetil (Experimental): Mycophenolate Mofetil 500 mg tablets of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Mycophenolate Mofetil
- Cellcept (Active Comparator): Cellcept 500 mg tablets of Roche Laboratories Inc.
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil 500 mg tablets
  Other Names: Cellcept

SUMMARY:
To compare the bioavailability and characterise the pharmacokinetic profile of the sponsor's test formulation with respect to the reference formulation Cellcept® 500 mg tablets, in healthy, adult, human male subjects under non-fasting conditions and to assess the bioequivalence.

DETAILED DESCRIPTION:
This was an open-label, balanced, randomized, two-treatment, two-period, two-sequence,single dose, crossover bioequivalence study in healthy, adult, human, male subjects under non-fasting conditions.92 healthy male adults were enrolled.A washout period of 07 days was maintained between the successive dosing days.One tablet containing mycophenolate mofetil 500 mg was administered orally with 240 mL water in sitting posture, after 30 minutes of serving of the high fat and high calorie breakfast in each period. This activity was followed by a mouth check to assess compliance to dosing. The subjects were not allowed to lie down for the first three hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males between 18-45 years of age (both inclusive) living in and around Mumbai city of western part of India.
2. Having a weight more than or equal to 50 Kg and having a Body Mass Index (BMI)between 18.5-24.9 (both inclusive), calculated as weight in kg / height in m2.
3. Having no significant diseases or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12-lead ECG and chest X-ray (postero-anterior view) recordings.
4. Able to comply with the study procedures, in the opinion of the Principal Investigator.
5. Able to give written consent for participation in the trial.

Exclusion Criteria:

1. Known hypersensitivity or idiosyncratic reaction to Mycophenolate Mofetil or any drug.
2. Any disease or condition which might compromise the haemopoietic, renal, hepatic,endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological,gastrointestinal or any other body system.
3. Ingestion of a medicine at any time with in 14 days before dosing in Period-I. In any such case subject selection will be at the discretion of the Principal Investigator /Medical Expert.
4. Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAID induced urticaria.
5. A recent history of alcoholism (<2 years) or of moderate (180 mL / day) alcohol use, or consumption of alcohol within 48 hours of receiving study medicine.
6. Smokers, who had a habit of smoking 10 or more than 10 cigarettes / day or could, not abstain from smoking during the study.
7. The presence of clinically significant abnormal laboratory values during screening.
8. Use of any recreational drugs or history of drug addiction or testing positive in pre-study urine drug scan.
9. History of psychiatric disorders.
10. A history of difficulty with donating blood.
11. Donation of blood (1 unit or 350 mL) within 90 days prior to receiving the first dose of the study medicine or during the study.

    Note: In case the blood loss was ≤ 200 mL, the subject was enrolled 60 days after blood donation.
12. A positive hepatitis screen including hepatitis B surface antigen and anti-HCV antibodies.
13. A positive test result for HIV antibody and / or syphilis.
14. The receipt of an investigational product or participation in a drug research study within a period of 90 days prior to the first dose of study medication. Elimination half-life of the study drug was taken into consideration for inclusion of the subject in the study.

    Note: If the subject had participated in a study in which blood loss was ≤ 200 mL, the subject was dosed 60 days after the collection of last sample in the previous study.
15. An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study medicine and throughout the subject's participation in the study. In any such case selection of the subject will be at the discretion of the Principal Investigator/Medical Expert.
16. Uric acid parameters at the time of screening are not within clinically acceptable range.
17. History of gout and renal calculi.
18. Sitting blood pressure less than 100/60 mm Hg at the time of screening.
19. Haemoglobin less than 13 gm/dL at the time of screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: T Gitanjali, MD, Principal Investigator — Lambda Therapeutic Research Ltd.
Locations (1):
- Lambda Therapeutic Research Ltd, Bodakdev, Ahmedabad, India